CLINICAL TRIAL: NCT03260049
Title: The Necessity and Optimal Time for Performing Pars Plana Vitrectomy in Acute Retinal Necrosis Patients
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shulin Liu, Dr., Chongqing Medical University
Other Study IDs: ChongqingMU-2
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Acute Retinal Necrosis
MeSH Terms: conditions — Retinal Necrosis Syndrome, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: there was no retinal detachment (RD) at the first visit. The group 1 patients were treated with systemic antiviral medications, as well as with intravitreal antiviral injections
- 2: there was no RD at the first visit. The group 2 patients were treated with systemic antiviral medications and PPV plus silicone oil tamponade and intravitreal injection.
  Interventions: Procedure: pars plana vitrectomy
- 3: there was RD at the first visit. The group 3 patients were treated with systemic antiviral medications and PPV plus silicone oil tamponade and intravitreal injection
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Procedure: pars plana vitrectomy — pars plana vitrectomy
  Other Names: systemic antiviral medications
  Groups: 2; 3

SUMMARY:
The records of patients who were diagnosed with ARN between April 2010 and February 2017 were analyzed.A retrospective review of the treatment options and outcomes of the these patients was performed.

ELIGIBILITY:
Inclusion Criteria:

* ARN was diagnosed according to the American Uveitis Society Diagnostic Criteria (1994)

Exclusion Criteria:

-

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARN patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
visual acuity | 1 year

SECONDARY OUTCOMES:
retinal detachement | 1 year

IPD SHARING:
Plan to Share IPD: No